CLINICAL TRIAL: NCT00002881
Title: PHASE III TRIAL OF ORCHIECTOMY/LHRH ANALOG + FLUTAMIDE + SURAMIN + HYDROCORTISONE VS ORCHIECTOMY/LHRH ANALOG + FLUTAMIDE IN PATIENTS WITH METASTATIC PROSTATE CANCER
Brief Title: Flutamide, Suramin, and Hydrocortisone in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065185; E-8892; CLB-E8892; SWOG-E8892
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2007-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin; Leuprolide; Suramin; Hydrocortisone; Orchiectomy

INTERVENTIONS:
Drug: flutamide
Drug: goserelin acetate
Drug: leuprolide acetate
Drug: suramin
Drug: therapeutic hydrocortisone
Procedure: orchiectomy

SUMMARY:
RATIONALE: Hormone therapy may be an effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to evaluate the effectiveness of treatment with flutamide and suramin with or without hydrocortisone in men who have metastatic or recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare time to progression and survival in patients with metastatic or recurrent adenocarcinoma of the prostate treated with orchiectomy or LHRH analogue (i.e. leuprolide or goserelin) plus flutamide with vs. without suramin and hydrocortisone. II. Compare these two treatments with respect to qualitative and quantitative toxic effects. III. Evaluate normalization of prostatic-specific antigen (PSA), duration of PSA response, and the use of PSA as a surrogate marker of tumor response in these patients. IV. Compare these two treatments with respect to quality of life and pain status.

OUTLINE: This is a randomized study. Patients are stratified by their choice of androgen suppression technique and by participating institution. Within 3 days after randomization, all patients receive daily flutamide. On day 4, patients undergo orchiectomy or begin monthly LHRH analogue therapy with leuprolide or goserelin. Patients randomized to receive suramin begin a 12-week course 8-25 days after orchiectomy/LHRH therapy. Hydrocortisone replacement therapy begins concomitantly with suramin and continues for at least 3 months after the completion of suramin treatment or until disease progression intervenes. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 800-1,000 patients will be entered within 3.25 to 4.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate that is stage D2 Measurable or evaluable disease required with at least one of the following: At least 7 bone lesions Visceral involvement No more than 50% replacement of liver by tumor No clinical suspicion of brain metastases No spinal cord compression

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 (ECOG 3 allowed if increase due only to pain) Life expectancy: At least 3 months Hematopoietic: (within 2 weeks prior to entry) WBC at least 3,000 AGC at least 1,500 Platelets at least 100,000 Hemoglobin at least 9.0 g/dL Hepatic: (within 2 weeks prior to entry) Bilirubin no greater than 2 times normal AST and ALT no greater than 2 times normal PT and PTT normal Albumin at least 3.0 g/dL Renal: Creatinine no greater than 2 mg/dL Creatinine clearance at least 60 mL/min BUN no greater than twice normal Cardiovascular: No myocardial infarction within 6 months No NYHA class III/IV status No history of thromboembolic or hemorrhagic cerebrovascular accident No disseminated intravascular coagulation No anticoagulant therapy (aspirin allowed for other uses) Other: No active bacterial infection No HIV or hepatitis B infection No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ cancer of any site

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biological response modifier therapy Chemotherapy: No prior chemotherapy (including suramin) Endocrine therapy: At least 1 year since any adjuvant or neoadjuvant hormone therapy No more than 4 months of therapy as part of initial prostate cancer therapy Prior finasteride for benign prostatic hypertrophy allowed No systemic steroids other than hydrocortisone (steroid inhalers allowed) Radiotherapy: At least 4 weeks since radiotherapy (90 days since strontium) Surgery: Recovered from prior surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-10; Primary Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison; Nancy A. Dawson, MD, Study Chair — Walter Reed Army Medical Center; A. O. Sartor, MD, Study Chair — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States